CLINICAL TRIAL: NCT01676454
Title: Determination of Serum Vasopressin Levels and Correlation With Life-threatening Complications in Adults With Severe Hemorrhagic Shock.
Brief Title: Serum Vasopressin Levels and Severe Hemorrhagic Shock
Status: Withdrawn | Type: Observational
Why Stopped: Study closed without enrollment .
Sponsor: Poudre Valley Health System (Other)
Responsible Party: Principal Investigator, Julie Dunn, M.D., Principal Investigator, Poudre Valley Health System
Other Study IDs: Vasopressin Study
Record Dates: First submitted 2012-08-21; First posted 2012-08-31 (Estimated); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Injury
Keywords: Vasopressin; Trauma; Injury
MeSH Terms: conditions — Wounds and Injuries; Diabetes Insipidus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vasopressin levels.: Cohort will consist of subjects with a minor injury or injuries defined as:
  1. no episodes of systolic blood pressure < 90 mmHg between occurrence of injury and admission;
  2. no blood transfusion requirement;
  3. base deficit < 5 mEq/L;
  4. no requirement for mechanical ventilation other than transiently during orthopedic surgery.

SUMMARY:
The purpose of this study is to determine if vasopressin is used up by the body during traumatic shock (severe low blood pressure due to trauma).

DETAILED DESCRIPTION:
For humans suffering trauma and severe hemorrhagic shock, no randomized controlled studies of the effect of exogenous vasopressin use exist, although case reports have suggested it may be of benefit. Even some moribund patients with "irreversible" shock survived severe hemorrhagic shock after administration of vasopressin. This suggests that at least some patients suffering severe trauma could benefit from AAVP administration. Recently, many clinicians and notable research consortiums have suggested that AVP shows promise for human resuscitation and have called for further human studies.

This is a prospective, single-center observational study designed to evaluate (1) whether vasopressin is depleted in severe, but not minor, trauma; and (2) the degree to which endogenous vasopressin levels predict the occurrence of ARDS, sepsis, or death. To test the first hypothesis, serum vasopressin levels (continuous independent variable) will be assessed at enrollment (time 0), 6, 12, 18, and 24 hours later, and correlated with the two levels of trauma (categorical dependent variable). To test the second hypothesis, serum vasopressin levels (now a continuous dependent variable) will be correlated with each of three outcomes-death, ARDS, and sepsis.

ELIGIBILITY:
Inclusion Criteria:

Patients with a minor injury or injuries, defined as:

1. no episodes of systolic blood pressure < 90 mmHg between occurrence of injury and admission;
2. no blood transfusion requirement;
3. base deficit < 5 mEq/L;
4. no requirement for mechanical ventilation other than transiently during orthopedic surgery.

Exclusion Criteria:

1. Pregnancy
2. corticosteroid use,
3. prisoners, and/or
4. head trauma as determined by computed tomography (head trauma may itself induce diabetes insipidus, a marker of pituitary damage and vasopressin deficiency), and/or
5. evidence of spinal cord injury (another cause of vasodilatory shock).

Patients will also be excluded if pre-hospital provider information cannot be obtained, or indicates that the trauma occurred more than one 1 hour prior to emergency department admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Medical Center of the Rockies with minor injuries.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Serum vasopressin levels. | 24 hours.
  6 mL's per blood draw for 5 timepoints=30 mL's total blood drawn.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Dunn, M.D., Principal Investigator — Poudre Valley Health System
Locations (1):
- Medical Center of the Rockies, Loveland, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: System website — http://pvhs.org/research